CLINICAL TRIAL: NCT03489447
Title: Mortality of Sepsis in Swedish Intensive Care Units 2008-2016
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/519
Record Dates: First submitted 2018-03-21; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis group: All adult (>= 18 years) patients with a diagnosis of sepsis included in the Swedish ICU Registry between 2008-01-01 and 2016-10-18
  Interventions: Other: ICU care
- Non-sepsis group: All adult (>=18 years) patients without a diagnosis of sepsis included in the Swedish ICU Registry between 2008-01-01 and 2016-10-18
  Interventions: Other: ICU care

INTERVENTIONS:
Other: ICU care — exposure to ICU treatment with or without diagnosed sepsis

SUMMARY:
A study of short and long term mortality in patients treated with or without a diagnosis of sepsis in Swedish intensive care units (ICU) 2008 - 2016. The cohort is characterized with regard to chronic comorbidity, severity of acute illness and demographic factors, and outcome is adjusted for these factors. Changes in mortality during the period are studied.

DETAILED DESCRIPTION:
All adult patients admitted to a general ICU included in the Swedish Intensive Care Registry (a majority of all ICUs in Sweden) between 2008-01-01 and 2016-10-18 are followed for one year and any deaths are registered. Data on illness severity scores, age, sex, admitting hospital and duration of ICU stay are recovered. Data are linked with the inpatient registry of the Swedish Board of Health and Welfare (Socialstyrelsen), and any discharge diagnoses from the last 5 years preceding ICU admission are recovered. These are used to assess chronic comorbidity.

Mortality, adjusted for severity of illness, comorbidity and patient factors, is studied and any changes over time during the inclusion period are assessed.

The data in the Swedish ICU Registry are entered by the treating ICU physicians and include severity of illness (Simplified Acute Physiology Score (SAPS)3), selected chronic comorbidity, sex and date of birth, ICU stay and selected interventions and complications. Relevant International Classification of Diseases (ICD)-10 diagnoses are required and assessment of the occurrence of severe sepsis or septic shock, during the inclusion period defined according to the American College of Chest Physicians/Society of Critical Care Medicine (ACCP/SCCM) (sepsis 2) criteria, is mandatory when entering data.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a Swedish general ICU (excluding specialized cardiothoracic, neurosurgical, pediatric and burns units) between 2008-01-01 and 2016-10-18
* Episode registered in Swedish Intensive Care Registry

Exclusion Criteria:

* Age < 18 years
* Readmission (only first episode during the period included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult general ICU patients included in the Swedish Intensive Care Registry 2008-01-01 to 2016-10-18.
Sampling Method: Non-Probability Sample
Enrollment: 252245 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
30 day mortality | From the day of ICU admission until death of any cause , whichever came first, assessed up to 30 days.
  mortality within 30 days after admission to ICU
90 day mortality | From the day of ICU admission until death of any cause, whichever came first, assessed up to day 90.
  mortality within 90 days after admission to ICU
365 day mortality | From the day of ICU admission until death of any cause , whichever came first, assessed up to day 365.
  mortality within 365 days after admission to ICU

SECONDARY OUTCOMES:
hospital mortality | From the day of ICU admission until death of any cause or day of hospital discharge, whichever came first, assessed up to day 365.
  mortality before discharge from hospital after admission to ICU
ICU length of stay | From the day of ICU admission until death of any cause or day of ICU discharge, whichever came first, assessed up to day 365.
hospital length of stay | From the day of ICU admission until death of any cause or day of hospital discharge , whichever came first, assessed up to day 365.

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Lipcsey, PhD, Principal Investigator — Uppsala University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strandberg G, Walther S, Agvald Ohman C, Lipcsey M. Mortality after Severe Sepsis and Septic Shock in Swedish Intensive Care Units 2008-2016-A nationwide observational study. Acta Anaesthesiol Scand. 2020 Aug;64(7):967-975. doi: 10.1111/aas.13587. Epub 2020 Apr 27. PMID 32232853

DOCUMENTS (1):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03489447/Prot_000.pdf